CLINICAL TRIAL: NCT03434093
Title: Modulation of the Parieto-frontal Communication
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left NIH
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 180054; 18-N-0054
Record Dates: First submitted 2018-02-14; First posted 2018-02-15 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Normal Physiology
Keywords: Paired Associative Stimulation (PAS); Functional Magnetic Resonance Imaging (fMRI); Electrical Field Modeling; Working Memory
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPC-DLPFC (Active Comparator): In this arm, the TMS paired-pulses will be first delivered over the posterior parietal cortex (PPC) and then over the dorsolateral prefrontal cortex (DLPFC)
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Behavioral: Working Memory Task
- DLPFC-PPC (Active Comparator): Arm Description: In this arm, the TMS paired-pulses will be first delivered over the over the dorsolateral prefrontal cortex (DLPFC) and then posterior parietal cortex (PPC)
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Behavioral: Working Memory Task

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Description: This will comprise single and repeated paired-pulses delivered over motor and non-motor areas.
Behavioral: Working Memory Task — This will consist in remembering an item presented 1 to 5 steps before the inquiry. This task will span the whole duration of the functional MRI acquisition.

SUMMARY:
Background:

Research shows that the parietal and prefrontal areas of the brain are involved in short-term memory. Researchers want to look at the effects of transcranial magnetic stimulation (TMS) of these areas on short-term memory and brain activity. They will use functional magnetic resonance imaging (fMRI) to look at brain activity.

Objective:

To look at the effects of TMS on brain pathways involved in memory.

Eligibility:

Healthy, right-handed adults ages 18-50

Design:

Participants will have 3 or 4 visits at least 1 week apart. They cannot drink alcohol for at least 48 hours before each visit.

The screening visit lasts about 1 (Omega) hours. It can be combined with the first testing visit. Screening includes:

* Medical history
* Physical exam
* Neurological exam
* Urine tests
* Questionnaires about being left or right handed and about their ability to imagine physical activities.

The first testing visit lasts about 1 (Omega) hours and includes an MRI. For the MRI, participants lie on a table that slides into a machine. They will lie still or perform simple memory tasks on a computer screen.

The second and third testing visits last about 3 hours. Participants will have:

* 2 MRIs
* TMS: A wire coil is held to the scalp. A brief electrical current passes through the coil to create a magnetic pulse that affects brain activity. They will perform simple memory tasks.
* EMG: Small electrodes are taped to the skin to record muscle activity while they rest.

After the study, participants will complete a questionnaire about any discomfort they experienced during the study.

...

DETAILED DESCRIPTION:
Objective: This study aims to identify whether repetitive dual-site transcranial magnetic stimulation (TMS) can modulate the functional connectivity between the parietal and dorso-lateral prefrontal cortices.

Study population: The study involves 26 healthy volunteers.

Design: This controlled study comprises 3 main visits for each subject: (1) a baseline, evaluation visit during which fMRI will be acquired during a visual short memory task along with diffusion tensor imaging and structural MRI; (2) a visit during which resting state fMRI (rsfMRI) will be acquired, followed by paired-associative stimulation (PAS) with pulses delivered over the parietal and then over the dorso-lateral prefrontal cortex, in order to induce a temporary plastic change in the interaction between the parietal and prefrontal cortices; the PAS will be followed by another rsfMRI and task fMRI; (3) a visit identical to #2 during which the PAS will be delivered with pulses in reverse order of previous visit.

Outcome measures: The effects of PAS will be quantified with rsfMRI and a short working memory task, considered as a proxy for complex motor and cognitive control.

* The primary outcome will be to investigate the resting state functional connectivity changes induced by each PAS intervention
* The secondary outcome #1 will be to evaluate the difference in visual angle error between sessions 2 and 3 in a working memory task during which the subjects will be asked to remember the position of a bar presented on the screen at different time intervals before the inquiry.
* The secondary outcome #2 will be to build an fMRI-DTI analysis pipeline for generation of TMS targets individually customized for each subject and a given task.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age between 18-50 years.
* Right-handed (handedness questionnaire will be part of the initial evaluation)
* Able to give informed consent.
* Have a normal neurological exam within the last year and MoCA>27
* Willing and able to abstain from alcohol for at least 48 hours prior to the study.
* Willing to not participate in other rTMS studies in the week preceding visits for the current protocol.

EXCLUSION CRITERIA:

-All participants must be able to undergo MRI and TMS, for which the MRI- and TMS-safety checklists will be part of the initial evaluation, and reconfirmed at the beginning of every visit. It will constitute as exclusion criteria if the participant:

* has metal in his/her body which would make having an MRI scan unsafe, such as pacemakers, stimulators, pumps, aneurysm clips, metallic prostheses, artificial heart valves, cochlear implants or shrapnel fragments, or if he/she was a welder or metal worker, since small metal fragments may be found in the eyes.
* is uncomfortable in small closed spaces (claustrophobia) so that he/she would feel uncomfortable in the MRI machine.
* is not able to lie comfortably on the back for up to 2 hours

has hearing loss.

--is pregnant.

* Self-reported consumption of >14 alcoholic drinks/week for a man and >7 alcoholic drinks/week for a woman.
* History of or current brain tumor, stroke, head trauma with loss of consciousness, epilepsy or seizures.
* Taking medications that act directly on the central nervous system such as anti-epileptics, anti-histamines, anti-parkinsonian medication, medication for insomnia, anti-depressants, anti-anxiety medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-03 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Resting state functional connectivity change induced by the paired associative stimulation | Study completion

SECONDARY OUTCOMES:
Difference in the visual angle error of a working memory task between the DLPFC-PCC and PPC-DLPFC paired associative stimulation | Study completion

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)

REFERENCES:
- [Background] Casula EP, Pellicciari MC, Picazio S, Caltagirone C, Koch G. Spike-timing-dependent plasticity in the human dorso-lateral prefrontal cortex. Neuroimage. 2016 Dec;143:204-213. doi: 10.1016/j.neuroimage.2016.08.060. Epub 2016 Aug 31. PMID 27591116
- [Background] Koch G, Ponzo V, Di Lorenzo F, Caltagirone C, Veniero D. Hebbian and anti-Hebbian spike-timing-dependent plasticity of human cortico-cortical connections. J Neurosci. 2013 Jun 5;33(23):9725-33. doi: 10.1523/JNEUROSCI.4988-12.2013. PMID 23739969
- [Background] Ma WJ, Husain M, Bays PM. Changing concepts of working memory. Nat Neurosci. 2014 Mar;17(3):347-56. doi: 10.1038/nn.3655. Epub 2014 Feb 25. PMID 24569831